CLINICAL TRIAL: NCT01687088
Title: Olfactory Acuity in Chronic Migraine: A Case-Control Study
Brief Title: Smell Sensitivity in Chronic Migraine: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MJM/Olfactory/002
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Migraine; Olfactory Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- chronic migraineurs: At least 8 migraine days per week and headache at least 15 days per month.
- controls: No significant headache or disability as defined by migraine disability scale.

SUMMARY:
Olfactory impairment is a common symptom of neurologic disorders and may be related to dopaminergic dysfunction. Studies show that patients with migraine show increased sensitivity to light and sound. In our previous study in episodic migraineurs, olfaction was similar to age and sex-matched controls outside of attacks, but lower during acute attacks.

The hypothesis is that olfactory function in chronic migraine (CM) will have mild impairment of olfaction at baseline but a more significant impairment during migraine or headache exacerbations.

The investigators have two objectives:

* To determine baseline olfactory acuity in subjects with CM and compare them to age and sex-matched controls
* To determine how olfaction changes during acute exacerbations of migraine in those with CM

To execute this study, the investigators will interview subjects and controls to ensure that they meet inclusion and exclusion criteria. After obtaining informed consent, subjects and controls will complete a questionnaire survey regarding their history or lack of history of headaches, smell sensitivity, osmophobia and current medication use and answer questions about attack frequency, location of headache, duration of disease, use of medication for pain, and disability. Both migraineurs and controls will take the University of Pennsylvania Smell Identification Test (UPSIT) in the office.

After the first visit, migraineurs and controls will self-administer the UPSIT at home. They will be required to return the second test to the Jefferson Headache Center.

The investigators will use analysis of variance (ANOVA) to determine variance in UPSIT scores between subjects and controls. To achieve a 90% power that the study will detect a statistically significant difference between the mean UPSIT scores at a two-sided 5 percent significance level, our sample size for both subjects and controls is 50.

DETAILED DESCRIPTION:
The investigators will interview subjects and controls to ensure that they meet inclusion criteria and do not meet exclusion criteria. After obtaining informed consent, subjects and controls will complete a questionnaire survey with the interviewer regarding their history of headaches, smell sensitivity, osmophobia and current medication use. Subjects will also answer questions about attack frequency, location of headache, duration of disease, use of medication for pain, and disability.

After completing the questionnaire survey, migraineurs and controls will take the University of Pennsylvania Smell Identification Test (UPSIT) in the office. During this visit we will demonstrate and give instructions on how to perform UPSIT at home.

After the first visit, migraineurs will self-administer the UPSIT during a migraine attack day at home. They will be required to mail or drop off the second test at the Jefferson Headache Center.

Age and sex matched controls will take the first UPSIT in the office. They will take second UPSIT 2 weeks later at home and call the Headache Center to notify the staff that they have completed the second UPSIT. They will be asked to mail or drop off the test at the Jefferson Headache Center.

The UPSIT is a standardized, validated test for olfaction. There are a total of 40 odorants, with four booklets each containing ten odorants. The stimuli are embedded in "scratch and sniff" microcapsules at the bottom of each page. Subjects must choose one answer among four possible answers for each odorant - a forced choice test. The validity and reliability of the UPSIT, as well as the basis for using these particular odorants, has been demonstrated in multiple studies. The tests kits will be supplied by Dr. Richard Doty at University of Pennsylvania.

The investigators will use analysis of variance (ANOVA) to determine variance in UPSIT scores between subjects and controls. We will also use ANOVA to examine differences based on subject characteristics, including attack frequency, duration of illness, osmophobia during attacks, and if odors trigger headaches. The investigators will also use Chi-square and the Wilcoxon rank sum test to determine categorical outcomes such as gender and statistical significance between groups.

To achieve a 90% power that the study will detect a statistically significant difference between the mean UPSIT scores at a two-sided 5 percent significance level, our sample size for both subjects and controls is 50. This is based on the assumption that the standard deviation of the response variable is 3 units. The investigator's assumptions about effect size are based on previous studies using the UPSIT to detect differences in subjects and controls in other neurologic disorders, such as schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over the age of 18 with Chronic Migraine (>15 headache days/month, at least 8 days meet criteria for migraine)

Exclusion Criteria:

* Subjects with sinus/nasal disease
* Subjects with a history of head trauma or degenerative disease
* Subjects who are decisionally impaired.
* Controls will be age and sex-matched with no history of migraine. They cannot have any disability from headache as determined by the MIDAS (Migraine Disability Assessment) questionnaire. Only controls with a MIDAS score of "0" (no disability) will be allowed in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects, over age 18 years who meet criteria for diagnosis of chronic migraine Controls will be age and sex-matched and will have no history of migraine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McNamara, MD, Principal Investigator — Thomas Jefferson University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Migraineurs | Controls
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Migraineurs | Controls | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Comparison of UPSIT Scores Between Subjects and Controls at Two Time Points
Description: Migraineurs and controls will take the University of Pennsylvania Smell Identification Test (UPSIT) in the office. The UPSIT test is a series of 40 questions and the score is the number of questions answered correctly. Each question is multiple choice and must be answered. The number of correct answers regarding the smells being experienced is the subjects score. The higher the score the better the sense of smell. This allows groups to be compared. In this study after the first visit, migraineurs will be given the UPSIT test without a headache and then they will self-administer the UPSIT during a migraine attack day at home.
  Age and sex matched controls will also take the first UPSIT in the office. They will take second UPSIT 2 weeks later at home.
Time Frame: Chronic migraineurs up to 12 months. Controls up to 2 weeks.
Measure: Mean (Standard Error); unit: UPSIT Score
Arm/Group | Chronic Migraineurs | Controls
Number analyzed (Participants) | 40 | 47
UPSIT Score
  First UPSIT Score | 34.5 (0.4) | 35.9 (0.1)
  Second UPSIT Score | 34.7 (0.4) | 36.1 (0.1)

ADVERSE EVENTS:
Arm/Group | Chronic Migraineurs | Controls
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No